CLINICAL TRIAL: NCT04542811
Title: Acupuncture For Preventing Of Attack Frequency And Improving Disability In Migraine Without Aura Patients
Brief Title: Acupuncture In Migraine Without Aura Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Cayir, Assoc. Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B.30.2.ATA.0.01.00/113
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Migraine Without Aura; Acupuncture
Keywords: migraine; acupuncture; MIDAS
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will take 12 sessions of acupuncture addition to their prophylaxis treatment. Acupuncture points will be bilateral LI-4, LI-11, ST-8, ST-44, SP-6, GB-1, GB-14, GB-20, LR-3, and GV-14, GV-20. Sterile and single-use stainless steel acupuncture needles measuring 0.25x25 mm will be inserted to a depth of 10 mm and be retained for 30 minute without any further stimulation. Acupuncture will be performed by an acupuncturist with an acupuncture practitioner licence from the Turkish Ministry of Health. Adverse events will be monitored for all acupuncture sessions.
  Interventions: Other: Acupuncture
- Control Group (No Intervention): Control group will take only their migraine prophylaxis treatment. Participants will followed-up 3 months.

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a complementary therapy modality which is used by needle inserted the specific points on the body.
  Arms: Intervention group

SUMMARY:
The investigators aimed to investigate the effect of acupuncture treatment on attack frequency, pain intensity, and disability in migraine without aura patients who receive prophylaxis treatment.

DETAILED DESCRIPTION:
Acupuncture is a Traditional Chinese Medicine method that has been used for 3000 years to control symptoms, treat illnesses, and relieve pain. Acupuncture is widely used in many countries today as a complementary therapy, especially in cases of chronic pain. Migraine is one of the diseases in which acupuncture treatment is commonly used. Studies conducted so far have focused more on the effect of acupuncture on pain intensity in patients with migraine. Data comparing the impact of acupuncture on both the attack frequency and disability in migraine are relatively scarce.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with migraine according to IHS (International Headache Association)
* Receiving migraine prophylaxis treatment
* Having more than four attacks per month/more than one attack per week
* Not having received acupuncture treatment before.

Exclusion Criteria:

* Being diagnosed with migraine with aura/secondary headache
* Having received acupuncture treatment for any reason within the last year
* Not giving consent for acupuncture treatment
* Having a fear of needles.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Monthly attack frequency | 3 months
  The participants will document the each migraine attack days in a month by pain free intervals of at least 48 hours.
Duration of attacks | 3 months
  Duration of the each migraine attack as hour
Pain severity | 3 months
  Pain severity during migraine attacks will be measured via visual analog scale (VAS). While 0 indicates no pain, 10 indicates the most severe pain imaginable.

SECONDARY OUTCOMES:
Disability | 3 months
  Disability will measured via a questionnaire which is an ordinary rating scale to assess the migraine related disability of a patient with migraine. Migraine Disability Assessment (MIDAS) will be used. Migraine Disability Assessment (MIDAS) questionnaire is an ordinary rating scale to assess the migraine related disability of a patient with migraine. It is based on responses to five questions about disability associated with headache in the last three months. MIDAS questionnaire has four point grading system. Scores ranging from 0 to 5 indicates Grade 1 (little or none disability), scores ranging from 6 to 10 indicates Grade 2 (mild disability), scores ranging from 11 to 20 indicates Grade 3 (moderate disability), and scores 21 or greater indicates Grade 4 (severe disability).

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Çayır, Study Director — Ataturk University
Locations (1):
- Rabia Rukiye Akinci, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No